CLINICAL TRIAL: NCT06858397
Title: An Open Label, Dose Range, Proof-of-Concept Study to Assess the Safety and Efficacy of HM15421/GC1134A in Patients With Fabry Disease
Brief Title: A proof-of Concept Study to Assess Safety and Tolerability of HM15421/GC1134A in Patients With Fabry Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC1134A_FD_P1201
Record Dates: First submitted 2025-02-19; First posted 2025-03-05 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Fabry Disesase

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Low dose
  Interventions: Drug: HM15421/GC1134A
- Cohort 2 (Experimental): Mid dose
  Interventions: Drug: HM15421/GC1134A
- Cohort 3 (Experimental): High dose
  Interventions: Drug: HM15421/GC1134A

INTERVENTIONS:
Drug: HM15421/GC1134A — SC

SUMMARY:
This Phase 1/2 first-in-human (FIH) study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of HM15421 in patients with FD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥ 18 years of age or age considered as adult in the respective country at the time of signing the informed consent.
2. Documented diagnosis of FD with clinical symptoms.
3. Females: historical genetic test results based on identification of pathogenic or likely pathogenic GLA variant of FD.
4. Males: Plasma and/or leucocyte alpha galactosidase activity (by activity assay) less than lower limit of normal (LLN in plasma=3.2 nmol/hr/mL, LLN in leucocytes=32 nmol/hr/mg/protein).
5. Patients who are naive or have not received FD therapy including investigational therapy for FD within the past 6 months prior to screening and have negative ADA testing at screening.
6. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
7. Plasma lyso-Gb3 levels greater than 1.5 times the upper limit of normal (ULN).
8. Male participants:

   * Male participants are eligible to participate if they agree to the following during the study treatment period:
   * Refrain from donating sperm,

   PLUS either:
   * Be abstinent from heterosexual intercourse with a woman of childbearing potential (WOCBP) as their preferred and usual lifestyle (abstinent on a longterm and persistent basis) and agree to remain abstinent, OR
   * Must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person,
   * In addition to male condom, use of highly effective method of contraception may be considered in WOCBP partners of male participants.
9. Female participants:

   * Female participants are eligible to participate if they are not pregnant or breastfeeding, and at least 1 of the following conditions applies:

     * Is not a WOCBP, OR
     * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, starting at least one menstrual cycle before first study drug administration and continuing for at least 30 days after the end of systemic exposure of the study drug and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study drug.
     * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study drug.
     * If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
   * Women whose postmenopausal status is recent, may perform additional follicle stimulating hormone (FSH) testing.

   Informed Consent
10. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Women who are pregnant, planning to become pregnant during the study, or are breast feeding.
2. History of dialysis or renal transplantation.
3. CKD stage ≥ 3.
4. History of acute kidney injury within 12 months prior to screening, including specific kidney diseases (eg, acute interstitial nephritis, acute glomerular and vasculitic renal diseases); non-specific conditions (eg, ischemia, toxic injury); as well as extrarenal pathology (eg, prerenal azotemia, and acute postrenal obstructive nephropathy).
5. Urine protein to creatinine ratio (UPCR) > 0.5 g/g and not treated with an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB).
6. Known history of hypersensitivity to any ingredient in the investigational product and to Gadolinium contrast agent that is not managed by the use of premedication.
7. Cardiovascular event (myocardial infarction, unstable angina) within 6 months before screening.
8. Congestive heart failure New York Heart Association (NYHA) Class IV
9. History of stroke.
10. Pacemaker or other contraindication for magnetic resonance imaging (MRI) scanning.
11. Angiotensin converting enzyme inhibitor or ARB therapy initiated or dose changed in the 4 weeks prior to screening.
12. Patients who received investigational gene therapy for FD.
13. Participation in other studies involving study drugs within 4 weeks prior to study entry and/or during study participation.
14. Participating in interventional study or using compassionate access product for FD. Participants who have participated in interventional trials for conditions not related to FD should be enrolled after the adequate wash out period is over, which is 5 half-lives or 30 days whichever is longer.
15. Presence of human immunodeficiency virus (HIV) and/or active (acute or chronic) hepatitis B and/or Hepatitis C infections.
16. Presence of any medical, emotional, behavioral, or psychological condition that, in the judgment of the Investigator and/or Medical Monitor, would interfere with the participant's compliance with the requirements of the study.
17. Participants who may have history of deliberate self-harm or suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidences and characteristics of adverse events | Up to 48 weeks

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | Up to 48 weeks
  PK parameter
Time to reach maximum serum concentration (Tmax) | Up to 48 weeks
  PK parameter
Trough serum concentration (Ctrough) | Up to 48 weeks
  PK parameter
Area under the concentration-time curve in one dosing interval (AUC0-tau) | Up to 48 weeks
  PK parameter
Terminal elimination half-life (t1/2) | Up to 48 weeks
  PK parameter
Apparent clearance at steady state (CLss/F) | Up to 48 weeks
  PK parameter
Apparant volume of distribution at steady state during the terminal phase (Vss/F) | Up to 48 weeks
  PK parameter
Plasma Lyso-Gb3 level | Up to 48 weeks
  PD parameter
Plasma Gb3 level | Up to 48 weeks
  PD parameter
Urine Lyso-Gb3 level | Up to 48 weeks
  PD Parameter
Urine Creatinine level | Up to 48 weeks
  PD parameter
Urine Albumin level | Up to 48 weeks
  PD parameter
Total Urine Protein Level | Up to 48 weeks
  PD parameter
Urine Protein to Creatinine Ratio | Up to 48 weeks
  PD parameter
Urine Albumin to Creatinine Ratio | Up to 48 weeks
  PD parameter
Change in eGFR | Up to 48 weeks
  PD parameter
Change in kidney Gb3 accumulation using the quantative Barisoni Lipid Inclusion Scoring System | Up to 48 weeks
  PD parameter

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - David Geffen School of Medicine UCLA, UCLA Health, Los Angeles, California
  - University of Kansas School of Medicine, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center Children's Hoispital of Pittsburgh, Pittsburgh, Pennsylvania
  - Lysosomal and Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Argentina (2):
  - Centro Medico IPAM, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
- South Korea (2):
  - Pusan National University Children's Hospital in Yangsan, Yangsan, Gyeongsangnam-do
  - Yonsei University, College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No